CLINICAL TRIAL: NCT06814106
Title: A Single- and Multiple-Dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-0616 in Healthy Chinese Adult Participants.
Brief Title: A Single- and Multiple-Dose Study of Enlicitide Chloride (MK-0616) in Healthy Chinese Adult Participants (MK 0616-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 0616-010; MK-0616-010 (Other: MSD)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Additional Roles Masked: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Enlicitide Chloride Panel A (Experimental): Period 1: Participants will receive a single dose of enlicitide chloride dose 1 or a single dose of placebo on Day 1 on an empty stomach (after a ≥8-hour overnight fast).
  Period 2: Participants will receive a single dose of enlicitide chloride dose 1 or a single dose of placebo on Day 1 on an empty stomach (after a ≥8-hour overnight fast) followed by a standard breakfast.
  Interventions: Drug: Enlicitide Chloride; Drug: Placebo
- Enlicitide Chloride Panel B (Experimental): Period 1: Participants will receive a single dose of enlicitide chloride dose 2 or a single dose of placebo on Day 1 on an empty stomach (after a ≥8-hour overnight fast).
  Period 2: Participants will receive a single dose of enlicitide chloride dose 3 or a single dose of placebo on Day 1 on an empty stomach (after a ≥8-hour overnight fast).
  Interventions: Drug: Enlicitide Chloride; Drug: Placebo
- Enlicitide Chloride Panel C (Experimental): Participants will receive enlicitide chloride dose 2 or placebo once daily for 14 days on an empty stomach (after a ≥8-hour overnight fast).
  Interventions: Drug: Enlicitide Chloride; Drug: Placebo

INTERVENTIONS:
Drug: Enlicitide Chloride — Oral Capsule
  Other Names: MK-0616
Drug: Placebo — Placebo oral capsule matching enlicitide chloride

SUMMARY:
The purpose of this study is to learn about the safety of enlicitide chloride and how well people tolerate it. Researchers also want to learn what happens to different amounts of enlicitide chloride in a healthy person's body over time.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to:

* Is in good health
* Has a body mass index ≥19.0 and ≤26.0 kg/m^2, inclusive

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

* Has a history of gastrointestinal disease
* Has a history of cancer (malignancy)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of Participants Who Discontinue the Study Treatment Due to an AE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention

SECONDARY OUTCOMES:
Panels A and B: Area Under the Concentration-Time Curve from 0 to Infinity (AUC0-inf) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the AUC0-inf of enlicitide chloride
Panels A and B: Area Under the Concentration-Time Curve from 0 to 24 Hours (AUC0-24) of Enlicitide Chloride | Predose and at designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of enlicitide chloride
Panels A and B: Area Under the Concentration-Time Curve from 0 to Last Measurable Concentration (AUC0-last) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the AUC0-last of enlicitide chloride
Panels A and B: Maximum Plasma Concentration (Cmax) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the Cmax of enlicitide chloride
Panels A and B: Time to Maximum Plasma Concentration (Tmax) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the Tmax of enlicitide chloride
Panels A and B: Concentration at 24 Hours Postdose (C24) of Enlicitide Chloride | 24 hours postdose
  Blood samples will be collected to determine the C24 of enlicitide chloride
Panels A and B: Apparent Terminal Half-Life (t1/2) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the apparent terminal t1/2 of enlicitide chloride
Panels A and B: Apparent Clearance (CL/F) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the CL/F of enlicitide chloride
Panels A and B: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Enlicitide Chloride | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the Vz/F of enlicitide chloride
Panels A and B: Percent of Reduction of Serum Low Density Lipoprotein Cholesterol (LDL-C) | Predose and at designated timepoints (up to 8 days postdose)
  Blood samples will be collected to determine the percent of reduction of serum LDL-C
Panel C: AUC0-24 of Enlicitide Chloride | Predose and at designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of enlicitide chloride
Panel C: Cmax of Enlicitide Chloride | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the Cmax of enlicitide chloride
Panel C: Tmax of Enlicitide Chloride | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the Tmax of enlicitide chloride
Panel C: C24 of Enlicitide Chloride | 24 hours postdose
  Blood samples will be collected to determine the C24 of enlicitide chloride
Panel C: Apparent Terminal t1/2 of Enlicitide Chloride | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the apparent terminal t/2 of enlicitide chloride
Panel C: CL/F of Enlicitide Chloride | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the CL/F of enlicitide chloride
Panel C: Vz/F of Enlicitide Chloride | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the Vz/F of enlicitide chloride
Panel C: Accumulation Ratio of Enlicitide Chloride | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the accumulation ratio of enlicitide chloride
Panel C: Percent of Reduction of Serum LDL-C | Predose and at designated timepoints (up to 14 days postdose)
  Blood samples will be collected to determine the percent of reduction of serum LDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharpe & Dohme LLC
Locations (1):
- Zhongshan Hospital,Fudan University-Dep. of Clinical Pharmacology (Site 0001), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com